CLINICAL TRIAL: NCT03766347
Title: Pediatric Neuromyelitis Optica Spectrum Disorder (NMOSD) 1 Year Observational Study
Brief Title: Pediatric NMOSD Observational Study
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Sean Pittock, Prinicpal Investigator, Mayo Clinic
Other Study IDs: 17-005618
Record Dates: First submitted 2018-12-04; First posted 2018-12-06 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Neuromyelitis Optica; NMO Spectrum Disorder
Keywords: Pediatric; Aquaporin-4; AQP4; NMOSD; NMO; Neuromyelitis Optica
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Neuromyelitis Optica: Participants under the age of 18 that are positive for Aquaporin-4 antibody.

SUMMARY:
This study is being done to develop a database of pediatric patients in order to study the cause, early detection and best treatment for neuromyelitis optica spectrum disorder (NMOSD) in pediatric patients.

DETAILED DESCRIPTION:
This study is being done to collect information on the natural history of NMOSD in pediatric AQP4-IgG seropositive patients. A major restriction in performing drug studies in pediatric patients with NMOSD is limited information on the course of the disease in these patients. Collecting clinical information over the course of a 1 year observational study would inform on the natural history of the disease in these patients. A repository of pediatric patients with rare diseases can increase knowledge on the natural history of the specific disease, assist in identifying appropriate patients fulfilling specified criteria for drug studies and potentially serve as a control group.

Timepoints: Baseline, 3mo, 6mo, 9mo, 12mo (+/- 1 mo for each time point).

Baseline data:

* Demographics [age/sex/ethnicity],
* Clinical presentation information including date of initial diagnosis,
* Clinical phenotype
* Immunotherapy used current and past,
* Family history of autoimmune diseases,
* Serological data results
* Radiologic data as available

Self-Report Assessments will be:

* Current impairment, as measured by the expanded disability status scale (EDSS) score self-reported using Ratzker (1997) EDSS Self Report form,
* Quality of life as measured by the EQ-5D and Varni's (1998) PedsQL over the phone/mail/email.

At follow-up visits 3mo, 6mo, 9mo, 12mo (+/- 1 mo for each time point):

* Attacks/relapses
* Any hospitalizations
* Confirm medications and update records if changes

Self-Report Assessments at follow-up will be:

* Current impairment, as measured by the EDSS score self-reported using Ratzker (1997) EDSS Self Report form,
* Quality of life as measured by the EQ-5D and PedsQL over the phone/mail/email.

ELIGIBILITY:
Inclusion Criteria:

* AQP4 positive
* Ability to give informed consent by patient or caregiver

Exclusion Criteria:

- Inability to complete required forms via phone, mail, or email.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Any pediatric patients that have tested positive for AQP4 antibody regardless of geographic location.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Time to relapse | One year.
  Relapse events of NMOSD defined by clinical worsening of neurological symptoms and treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sean J Pittock, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials